CLINICAL TRIAL: NCT01126905
Title: A Local Pilot Evaluation of Laboratory Monitoring of Renal Patients on Erythropoietin and /or Iron Therapy Using Mean Reticulated Haemoglobin Equivalent (RetHe) and Their Response to Therapy
Brief Title: Mean Reticulated Haemoglobin (Hb) Content (RetHe) Analysis of Renal Patients
Status: Completed | Type: Observational
Sponsor: University of Ulster (Other)
Collaborators: NHS Fife (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2010FAL1
Record Dates: First submitted 2010-05-19; First posted 2010-05-20 (Estimated); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: End-Stage Renal Failure; Functional Iron Deficiency
Keywords: Reticulated Haemoglobin Equivalent; Functional Iron Deficiency; Response to therapy; Iron deficiency
MeSH Terms: conditions — Kidney Failure, Chronic; Iron Deficiencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Anaemia is a common complication of Chronic Kidney Disease (CKD) the management of which has been aided by the use of synthetic recombinant human erythropoietin therapy (r-HuEPO). This red cell stimulating agent creates the further complication of Functional Iron Deficiency (FID) where, despite normal iron stores, patients fail to respond to therapy as they do not possess enough available iron to meet the demand of increased red cell production. Effective response to r-HuEPO therapy depends on an appropriate monitoring of 'available' iron levels.

Previous research into the clinical utility of testing for reticulated haemoglobin concentrations (Ret He) instead of Serum Ferritin and Transferrin Saturation analysis has indicated an advantage as an iron deficient prognostic marker however, further knowledge is required on the use of this new laboratory test (RetHe) to predict Functional Iron Deficiency (FID) level and to study it's relationship with responses to therapy.

This proposed study aims to estimate a local working Normal (non deficient) and Iron Deficient Reticulated Haemoglobin Content (RET He) reference range from surplus anonamous samples. Routine monthly blood samples from Pre Dialysis and Haemodialysis patients will be used to evaluate the sensitivity and specificity of the RET He test compared to current laboratory tests and investigate its predictive ability for Functional Iron Deficiency in these patients.

Studying , measuring and statistically analysing the change in the RET He parameters in Haemodialysis and Pre Dialysis patients over 3 months will look for evidence of a direct relationship between RET He values and the patients response to therapy. The data will be used to provide a predictive picture of what levels of RET He indicate Functional Iron Deficiency.

The introduction of this test (RetHe) may provide clinicians with a one sample/one test control over iron therapies and ensure the patient gets the most benefit from erythropoietin therapy.

DETAILED DESCRIPTION:
Reference Range Testing for new test RET-He will be performed on excess blood available on randomly selected anonamised samples obtained from the daily workload of the laboratory once all the clinically requested analysis has been completed.

100 samples (50 men / 50 women)determined to have normal parameters(as defined by Dacie et al, 10th Edition) and 100 samples (50 men / 50 women)determined to be iron deficient (as defined by Dacie et al, 10th Edition)will be processed for new test parameter (RetHe) under a coded number to ensure no identifying data is recorded. The samples will be archived and and held within the lab for 24 hours prior to routine disposal in accordance with NHS Fife Waste Management Policy.The data will be analysed using a paired t test to determine significant differences and reference range inferred inferred.

Evaluation of sensitivity / specificity of new Ret He test in determinimg iron deficiency and functional iron deficiency and it's response to terapy will be tested using Haemodialysis and Pre-Dialysis Patient Samples (~180 Haemodialysis Patients and ~250 Pre Dialysis Patients)that are obtained during their normal renal unit / clinic appointments.

All consenting NHS Fife Haemodialysis /Pre Dialysis patients will be allocated a 'Subject Identification Number' as part of this study (which will be noted at the top of their Consent Form). This number will be used by the Student Investigator to generate a confidential Coding Key which will be kept separate from data information and secure uner an NHS password protected computer. This will ensure care of personal information and will be used through-out the study by the student investigator to record all generated data.

Patients will be grouped into categories such as Dialysis / Pre Dialysis on a coded SPSS (statistical software) file.

All consenting patients will attend their routine scheduled Renal Clinic appointments as normal (no additional appointments are necessary for this pilot study)and their response to therapy will be observed using the new RetHe test parameter compared to existing laboratory tests utlised (FBC,Ferritin and Transferrin Saturation Levels)

Haemodialysis Patients - June 2010, July 2010*, August 2010

(* NB: In July 2010 Haemodialysis patients are scheduled to have their Ferritin and Transferrin Saturation Levels checked and therfore no additional sample will be required)

1. Routine venesection of EDTA (purple topped) sample for Full Blood Count (FBC) Test
2. Routine venesection of Clotted (yellow topped) sample for Biochemistry Analysis
3. Additional venesection of extra yellow topped sample for non routine Ferritin Test(*usually scheduled every 3 months- routine date due: July 2010)
4. Renal Unit Staff label samples and complete request form:

   Haematology section ticked for: FBC (as normal routine) , Retics (to allow addition of new Ret He test to FBC analysis) and Ferritin (additional request in June and August)

   Biochemistry section ticked for : All routinely requested Biochemistry tests (such as Urea and Electrolytes) plus additional request for Transferrin Saturation Levels (in June and August)
5. Sample and Requests sent to Fife Area Lab for Analysis

   The project will be carried out within NHS Fife Area Laboratory Haematology Department and will involve the use of NHS premises, facilities and staff.
6. Request checked at Laboratory Central Reception (sample and request form labelled with unique positive barcode identification)
7. Request Forms sent to central request entry and samples delivered to appropriate laboratories
8. FBC samples checked prior to analysis to check request details entered into Laboratory Host Computer System
9. FBC sample loaded onto Sysmex XE2100 Haematology Analyser for testing
10. Bidirectional Computer Link between Laboratory Host Computer System and Analyser ensures sample tested for FBC and additionally requested RETIC (reticulocyte analysis)
11. Sysmex XE2100 automatically analyses sample for Red Blood Cell Indices and additionally uses fluorescent polymethine dye to stain for RNA/DNA content of reticulated cells (early red blood cell precursors). The analyser uses inbuilt Flow Cytometry and measures forward scatter to separate cells by size (this is reported as RBC-Y and RET-Y)
12. Sysmex XE2100 RETIC Master software (recently upgraded packaged loaded onto NHS Fife Analysers)uses an algorithm (RET-He = 5.5569e 0.001RET-Y) to convert RET-Y into a reportable mean reticulocyte haemoglobin content (RET He) which is expressed in picograms.
13. The sample once analysed is removed from the analyser and the results are either autovalidated and archived (if results are within normal range) or held for validation by a NHS Fife qualified Biomedical Scientist.
14. The routinely requested FBC results are available for clinicians within same timescale as normal (no delay due to additional RetHe analysis)
15. The sample is archived under their unique identifying barcode numbers and held within the lab for 24 hours prior to routine disposal in accordance with NHS Fife Waste Management Policy.
16. The new RetHe value will be held on Sysmex XE2100 analyser (not activated as a reportable test to NHS Fife Biomedical Scientists or clinical staff.)
17. The Student Investigator will (on same day as analysis) retrospectively generate a Renal Unit worklist from the Laboratory Host Computer System which will indicate: how many samples received, barcode numbers, names of patients.
18. The Student Investigator will (on same day as analysis) retrospectively use the generated worklist to search the Sysmex XE2100 analysers for Ret-He test results and the host computer system for results of Ferritin and Transferrin Saturation Levels.
19. The barcode number of the patient and their test results will initially be recorded in the student investigators laboratory handbook (the generated worklist will be discarded into NHS Fife Confidential Waste)
20. The student investigator will record the test values into a coded SPSS (statistical software) file for appropriate analysis.
21. The investigator will retrospectively match the test data with therapy regime data provided by the Renal Unit (monthly meetings)

Pre Dialysis Patients: June 2010, July 2010, August 2010

(NB: Pre Dialysis Patients are tested 3 monthly so over period of study should get a baseline sample from each consenting patient. Only those patients who are considered iron replete and are placed on 5 week course of iron therpay will be further tested at their follow-up appointments in order to measure response to therapy)

1. Routine venesection of EDTA (purple topped) sample for Full Blood Count (FBC) Test, clotted (yellow topped) for Ferritin and clotted (yellow topped)sample for Transferrin Saturation Levels
2. Renal Unit Staff label samples and complete request form:

   Haematology section ticked for: FBC (as normal routine) , Retics (to allow addition of new Ret He test to FBC analysis) and Ferritin (routine request)

   Biochemistry section ticked for : All routinely requested Biochemistry tests (such as Urea and Electrolytes) plus routine request for Transferrin Saturation Levels
3. Sample and Requests sent to Fife Area Lab for Analysis

The project will be carried out within NHS Fife Area Laboratory Haematology Department and will involve the use of NHS premises, facilities and staff (same process as points 6 - 21 above)

ELIGIBILITY:
Inclusion Criteria:

* Two groups of random routine anonamised blood samples (for use in determinimg a local normal range for the Reticulated Haemoglobin Content [RetHe])will be included in the study:

Normal red blood cell (RBC) Indices (Hb , Haematocrit, Mean Cell Volume ande Mean Cell Haemoglobin Content) ; an attempt will be made to select an equal mixture of men / women and an appropriate age spread to provide a valid control range for the group of test subjects (renal patients) The student Investigator will ask Haematology staff to record minimum details of iron deficient patients and "normal" test results noted at routine validation [positive identification number (barcode)/ age / sex] - these samples will be coded and additionally analysed for RetHe test.

Exclusion Criteria:

* All renal patient who have had surgery and / or a Blood Transfusion OR bleeding episodes within the last month prior to the study are excluded as this would interfere with red cell parameters.

All patients < 16 years and >85 years are excluded from the study.

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Renal Patients requested to participate in study (consent required)
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2010-06; Primary Completion 2010-10-07 (Actual); Study Completion 2010-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Robson, Study Director — NHS Fife Laboraories; PAMELA MARKS, BSc Hons., Principal Investigator — NHS Fife Area Laboratory